CLINICAL TRIAL: NCT02920515
Title: Multi-site Study of Comprehensive Treatment for Children Precocious Puberty
Brief Title: Study of Comprehensive Diagnosis and Treatment for Children Precocious Puberty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other); Xin Hua Hospital (Other)
Responsible Party: Principal Investigator, WeiWang, professor, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12411950400
Record Dates: First submitted 2016-08-16; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Central Precocious Puberty
Keywords: epidemiology; treatment; molecular pathological mechanism; environmental disrupting chemicals
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GnRHa(Triptorlin or Leuprorelin) (Experimental): Triptorlin or Leuprelin 100ug/kg per 28 days
  Interventions: Drug: Triptorlin or Leuprorelin
- Traditional Chinese Medicines (Active Comparator): Zhibo dihuang pills: 8 tablets twice a day by mouth for 6 months and Dabu ying pills: 6g twice a day by mouth for 6 months
  Interventions: Drug: Zhibo dihuang pills; Drug: Dabu ying pills
- blank group (No Intervention): without therapy

INTERVENTIONS:
Drug: Triptorlin or Leuprorelin — Gonadotrophin releasing hormone agonists (GnRHa)
  Other Names: Triptorlin; Leuprorelin
  Arms: GnRHa(Triptorlin or Leuprorelin)
Drug: Zhibo dihuang pills — Traditional Chinese Medicine
  Arms: Traditional Chinese Medicines
Drug: Dabu ying pills — Traditional Chinese Medicine
  Arms: Traditional Chinese Medicines

SUMMARY:
This is a prospective, multicentric, comparative, non-randomized interventional study in which subjects diagnosed with central precocious puberty (CPP) and early puberty (EP) were treated for 6 months to compare the effect with GnRHa and traditional Chinese medicines.

DETAILED DESCRIPTION:
740 girls with CPP and EP participated in this study, all participates were divided into GnRHa group, traditional chinese medicines group and blank group. After at least six months therapy with GnRHa or traditional Chinese medicines, the investigators compare clinical parameters, sex hormone, bone age and ovarian ultrasound in three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Premature appearance of secondary sexual characteristics: girls present with development of secondary sexual characteristics before 8, with breast induration as the earliest manifestation.
2. Accelerated linear growth: the annual growth rate is higher than normal.
3. Advanced bone age: the bone age is 1 or years more than the actual age
4. Enlargement of sexual glands: B-mode ultrasonography of pelvic cavity indicates the volumes of the uterus and ovaries have increased, and multiple ovarian follicles with a diameter>4mm can be found in ovaries;
5. HPGA functions have been primed; serum gonadotropin and sexual hormone levels reach pubertal values.
6. Subjects should be willing and able to follow the study protocol during the study period.
7. Subjects should submit their parents' or guardians' written informed consent before initiation of the study procedure with non-normal medical care. They should understand that subjects or their parents/guardians may withdraw the consent at any time without impairing future medical care. If the child is old enough to read and write, she should submit a separate consent form.

Exclusion Criteria:

1. Patients with central nervous system diseases and thyroid diseases;
2. Patients with CHA-induced precocious puberty;
3. Patients with poor compliance.

Ages: 2 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 740 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Comparisons of the height SDS'changes between GnRHa group and traditional chinese medicines group in 6 months. | 6 months
  The change levels of height SDS in the GnRHa group (n=202) is lower than in the traditional chinese medicines group (n=155) ,(P<0.05).

SECONDARY OUTCOMES:
Comparisons of the breast stages'changes between GnRHa group and traditional chinese medicines group in 6 months. | 6 months
  The change levels of breast stages in the GnRHa group (n=181) is lower than in the traditional chinese medicines group (n=148) ,(P<0.05).

OTHER OUTCOMES:
Comparisons of the BA/CA ratio'changes between GnRHa group and traditional chinese medicines group in 6 months. | 6 months
  The change levels of BA/CA ratio in the GnRHa group (n=152) is lower than in the traditional chinese medicines group (n=86) ,(P<0.05).
Comparisons of the sex hormone'changes between GnRHa group and traditional chinese medicines group in 6 months. | 6 months
  The change levels of sex hormone(LH,FSH and E2) in the GnRHa group (n=164) is lower than in the traditional chinese medicines group (n=94) ,(P<0.05).
Comparisons of the uterine volume'changes between GnRHa group and traditional chinese medicines group in 6 months. | 6 months
  The change levels of uterine volume in the GnRHa group (n=157) is lower than in the traditional chinese medicines group (n=91) ,(P<0.05).
Comparisons of the ovarian volume'changes between GnRHa group and traditional chinese medicines group in 6 months. | 6 months
  The change levels of ovarian volume in the GnRHa group (n=152) is lower than in the traditional chinese medicines group (n=88) ,(P<0.05).

CONTACTS AND LOCATIONS:
Overall Officials: Pin Li, Dr, Principal Investigator — Shanghai Children's Hospital; Xuefan Gu, Dr, Principal Investigator — Xin Hua Hospital; Xiaodong Huang, Dr, Principal Investigator — Shanghai children's medicial Center; Fan Jiang, Dr, Principal Investigator — Shanghai children's medicial Center

IPD SHARING:
Plan to Share IPD: Yes